CLINICAL TRIAL: NCT04433065
Title: The Early Feasibility Study of the Transcatheter Tricuspid Valve Replacement System Transfemoral System
Brief Title: TTVR Early Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT20009TMV003
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Primary Cohort (Experimental): Device: Intrepid TTVR System
  Interventions: Device: Intrepid™ TTVR System

INTERVENTIONS:
Device: Intrepid™ TTVR System — Device: Intrepid™ TTVR System

SUMMARY:
The objective of this early feasibility study is to gain early clinical insight into the performance of the Intrepid transcatheter tricuspid valve replacement (TTVR) system intended for transfemoral access to deliver a self-expanding bioprosthetic valve within the tricuspid valve.

DETAILED DESCRIPTION:
Multi-center, prospective, non-randomized, investigational, and pre-market.

ELIGIBILITY:
Inclusion Criteria:

* Heart Team agrees that patient is deemed symptomatic despite medical therapy (including obligatory diuretic) and a candidate for bioprosthetic tricuspid valve replacement
* Subject is at an intermediate or greater estimated risk of mortality with tricuspid valve surgery as determined by the local Heart Team
* Subjects with severe symptomatic primary and / or secondary tricuspid regurgitation determined by the Echocardiography Core Lab assessment of a qualifying transthoracic echocardiogram (TTE) and transesophageal echocardiogram (TEE)
* New York Heart Association (NYHA) Function Class II or greater
* Subject anatomically suitable for the Intrepid TTVR delivery system including transfemoral access
* Subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits
* Subject meets the legal minimum age to provide informed consent based on local regulatory requirements

Exclusion Criteria:

* Estimated life expectancy of less than 24 months due to associated non-cardiac co-morbid conditions
* Anatomic contraindications for Intrepid™ TTVR (e.g., annular dimensions)
* Evidence of intracardiac mass, inferior vena cava, or femoral venous mass or thrombus
* Implanted with venous stents (iliac and/or femoral) or inferior vena cava (IVC) filter or congenital abnormalities of the IVC that would preclude ability for transfemoral access of delivery system
* Echocardiographic evidence of severe right ventricular dysfunction
* Left ventricular ejection fraction (LVEF) <30 as measured by resting echocardiogram within 30 days of the Index Procedure
* Need for emergent or urgent surgery
* Untreated clinically significant coronary artery disease requiring revascularization
* Carcinoid tricuspid regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2031-07-30 (Estimated)

PRIMARY OUTCOMES:
Rate of implant or delivery related serious adverse events | Through 30 days post-procedure
  Rate of implant or delivery related serious adverse events

SECONDARY OUTCOMES:
Successful access, delivery of implant, and retrieval of the delivery system assessed by definitions per Mitral Valve Academic Research Consortium (MVARC) | During Procedure
  For procedural success to be present, device success must have been achieved without major clinical complications as detailed per clinical trial design principles and endpoint definitions for transcatheter mitral valve repair and replacement (part 2: endpoint definitions)
Change in TR Grade from baseline | Through 30 days post-procedure
  Change in TR Grade from baseline
Rate of no significant TV stenosis | Through 30 days post-procedure
  Rate of no significant TV stenosis
Change in NYHA Class from baseline | Through 30 days post-procedure
  Change in NYHA Class from baseline

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Hartford Hospital, Hartford, Connecticut
  - Emory University Hospital Midtown, Atlanta, Georgia
  - University of Michigan Health System - University Hospital, Ann Arbor, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Providence Saint Patrick Hospital, Missoula, Montana
  - The Mount Sinai Hospital, New York, New York
  - New York-Presbyterian Hospital Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - UPMC Pinnacle Harrisburg Campus, Harrisburg, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - Aurora Saint Lukes Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No